CLINICAL TRIAL: NCT00256633
Title: CSP #465C - Fatty Acid Binding Protein 2 (FABP2) Ancillary Proposal
Brief Title: Fatty Acid Binding Protein 2 (FABP2) Ancillary Proposal
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 465C; 9066 (Other Grant/Funding Number: Minnesota Medical Foundataion)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Blood draws of DNA samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2.

SUMMARY:
TITLE: CSP 465-C, Fatty Acid Binding protein 2 (FABP2) ancillary proposal to CSP# 465 Glycemic Control and Complications in Diabetes Mellitus Type 2.

Angeliki Georgopoulos, M.D. Carlos Abraira M.D. William Duckworth M.D.

Fatty acid binding protein 2 (FABP2) is involved in the transport of long chain fatty acids across the intestinal epithelium. A common (40-45%) polymorphism of FABP2 gene (codon 54 Threonine for Alanine) results in increased intestinal fatty acid absorption and triglyceride secretion (Baier et al J Clin Invest 95:1281-87, 1995; Baier et al J Biol Chem 271: 10892-10896,1996). We have found (JCEM 85:3155-60, 2000) that in patients with type 2 diabetes, the codon 54 polymorphism of the FABP2 results in fasting and postprandial hypertriglyceridemia. Since hypertriglyceridemia is a risk factor for atherosclerosis in type 2 diabetes and it is part of the insulin resistance syndrome, the objective of this ancillary study would be to screen the participants of the CSP# 465 study for the polymorphism and assess a) whether those carrying the polymorphism respond differently to the various treatment modalities and b) whether they develop more cardiovascular events compared to the ones lacking the polymorphism. There is one study that suggests an association of the polymorphism with a history of parental stroke (JCEM 85:2801-4, 2000).

The only additional request from the study participants will be to agree to the collection of a blood sample to be used for DNA isolation and screening for the polymorphism. No additional funds are requested. If this polymorphism proves to be a predictor of either the response to a specific treatment modality or of the risk to macro-vascular complications, it will be very easy to screen for it and target our treatment modalities appropriately.

DETAILED DESCRIPTION:
Primary Hypothesis:

Secondary Hypotheses:

Primary Outcomes: Major cardiovascular events

Study Abstract:

TITLE: CSP 465-C, Fatty Acid Binding protein 2 (FABP2) ancillary proposal to CSP# 465 Glycemic Control and Complications in Diabetes Mellitus Type 2.

Angeliki Georgopoulos, M.D. Carlos Abraira M.D. William Duckworth M.D.

Fatty acid binding protein 2 (FABP2) is involved in the transport of long chain fatty acids across the intestinal epithelium. A common (40-45%) polymorphism of FABP2 gene (codon 54 Threonine for Alanine) results in increased intestinal fatty acid absorption and triglyceride secretion (Baier et al J Clin Invest 95:1281-87, 1995; Baier et al J Biol Chem 271: 10892-10896,1996). We have found (JCEM 85:3155-60, 2000) that in patients with type 2 diabetes, the codon 54 polymorphism of the FABP2 results in fasting and postprandial hypertriglyceridemia. Since hypertriglyceridemia is a risk factor for atherosclerosis in type 2 diabetes and it is part of the insulin resistance syndrome, the objective of this ancillary study would be to screen the participants of the CSP# 465 study for the polymorphism and assess a) whether those carrying the polymorphism respond differently to the various treatment modalities and b) whether they develop more cardiovascular events compared to the ones lacking the polymorphism. There is one study that suggests an association of the polymorphism with a history of parental stroke (JCEM 85:2801-4, 2000).

The only additional request from the study participants will be to agree to the collection of a blood sample to be used for DNA isolation and screening for the polymorphism. No additional funds are requested. If this polymorphism proves to be a predictor of either the response to a specific treatment modality or of the risk to macro-vascular complications, it will be very easy to screen for it and target our treatment modalities appropriately.

The data was not analyzed therefore there will be no results for this record/study.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 DM who are no longer responsive to maximum dose of one or more oral agents.

Exclusion Criteria:

Patients not registered in the VADT.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study of patients who are enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2.
Sampling Method: Non-Probability Sample
Enrollment: 874 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be to determine if DNA characteristics are associated with CV risk in type 2 diabetes mellitus. | End of study.

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Georgopoulos, MD, Study Chair — Minneapolis Veterans Affairs Medical Center; Carlos Abraira, MD, Study Chair — Miami VA Healthcare System, Miami, FL; William Duckworth, MD, Study Chair — Carl T. Hayden VA Medical Center
Locations (16):
- United States (15):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Central California Health Care System, Fresno, Fresno, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, Miami, Miami, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Omaha, Omaha, Nebraska
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Nashville, Tennessee
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Medical Center, Salem VA, Salem, Virginia
- VA Medical Center, San Juan, San Juan, Puerto Rico